CLINICAL TRIAL: NCT06871462
Title: Implementation Strategies for Self-Measured Blood Pressure Monitoring in Racially and Ethnically Diverse Populations
Acronym: INSPIRED
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); Beth Israel Deaconess Medical Center (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-42092; R18HS029817 (AHRQ)
Record Dates: First submitted 2025-03-04; First posted 2025-03-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Blood Pressure Monitoring, Home; Hypertension
Keywords: INSPIRED
MeSH Terms: conditions — Hypertension; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Intensity (Usual Care) (Active Comparator): Patient level: training on how to use a blood pressure (BP) monitor and online patient portal (ex. MyChart), receive reminders to take their BP at home, receive educational messages, and access to language-concordant educational materials.
  Clinic level: training on standardized workflows and EHR tools, audit and feedback
  Interventions: Behavioral: BP monitor use training and app training; Behavioral: Online patient portal enrollment and training; Behavioral: SMS reminders to take blood pressure; Behavioral: Education about self-management of hypertension
- High-Intensity (Experimental): Patient level: In addition to the Low-Intensity Arm strategies, patients will be asked to attend four educational group sessions with other trial patients. Patients will also be asked to involve support persons in their hypertension management. The educational messages that patients receive will also explicitly encourage involvement of a support person.
  Clinic level: training on standardized workflows and EHR tools, audit and feedback
  Interventions: Behavioral: BP monitor use training and app training; Behavioral: Online patient portal enrollment and training; Behavioral: SMS reminders to take blood pressure; Behavioral: Education about self-management of hypertension; Behavioral: Educational text messages that encourage seeking support from a support person; Behavioral: Involvement of caregiver or support person; Behavioral: Group classes

INTERVENTIONS:
Behavioral: BP monitor use training and app training — Patients will be taught how to use a BP monitor, along with the accompanying mobile app to view their readings.
Behavioral: Online patient portal enrollment and training — Patients will receive training on how to use an online patient portal. If they are not yet enrolled in an online patient portal and would like to be, they will also be enrolled into one.
Behavioral: SMS reminders to take blood pressure — Patients will receive reminders via SMS to take their blood pressure.
Behavioral: Education about self-management of hypertension — One-time training with action planning, access to website with language concordant patient education, and educational text messages
Behavioral: Educational text messages that encourage seeking support from a support person — Educational text messages about behavioral changes that explicitly encourage seeking support from a support person
  Arms: High-Intensity
Behavioral: Involvement of caregiver or support person — Patients will be asked to involve a caregiver or support person for all activities above, including patient portal proxy access.
  Arms: High-Intensity
Behavioral: Group classes — Patients will be asked to attend in-person or online group education classes on hypertension management
  Arms: High-Intensity

SUMMARY:
This clinical trial aims to assess the impact of patient-focused and clinical-focused implementation strategies on blood pressure control. The investigators will assess the costs of these strategies and how effective they were at safely and equitably increasing home blood pressure monitoring.

DETAILED DESCRIPTION:
This study will focus on assessing implementation strategies to increase adoption of self-monitored blood pressure (SMBP) monitoring among low-income, culturally and linguistically diverse patients with hypertension in an urban safety net. The investigators propose a hybrid type 1 effectiveness-implementation trial of implementation strategies to increase use of SMBP monitoring with clinical support in an urban safety net system. 330 patients will be randomized to a low-intensity vs high-intensity implementation strategy for SMBP monitoring. The low-intensity strategy will replicate frequently used implementation efforts (provision of BP monitor with training on using a monitor) while the high-intensity strategy will address additional factors identified in prior work (e.g., digital literacy, social support). In six adult primary clinics, the investigators will concurrently provide a stepped-wedge clinic-level implementation strategy (clinical champions, electronic health record [EHR] tools) to increase provision of clinical support for SMBP data. To guide dissemination in other under-resourced settings, an economic evaluation will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old/order
* Any sex or gender
* Any race or ethnicity
* Must be receiving primary care at any of the six enrolled clinics
* Have uncontrolled hypertension (BP >=140/90 mmHg at any two encounters in the previous 18 months, including the most recent encounter prior to enrollment)
* Can read and write English, Spanish, or Cantonese
* Be able to provide consent
* Must own a cell phone that receives SMS or text messages

Exclusion Criteria:

* Those with conditions that might complicate remote BP monitoring:

  * Pregnancy (and 12 months postpartum)
  * Acute myocardial infarction or stroke in the last 12 months
  * End-stage renal disease on dialysis
  * Stage D heart failure
  * Active treatment for cancer (except for nonmelanoma skin cancers)
  * Pacemaker use
* Those with dementia, in hospice care, or with serious behavioral health conditions impeding participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in clinic systolic BP | Baseline, 12 months, 18 months
BP Control | Monthly (-6 to 18 months)
  Clinic patients with EHR recorded BP < 140/90

SECONDARY OUTCOMES:
BP Control | Baseline, 12 months, 18 months
  Enrolled participants with controlled BP based on (a) clinic BP values; (b) home BP values
Home Systolic BP (SBP) | Baseline, 12 months, 18 months
  Home SBP for enrolled participants
Patient Adoption | 12 months
  Number of SMBP values per participant
Clinic adoption | Monthly (-6 to 18 months)
  Clinic patients with EHR documented patient reported BP
Reach | 12 months
  Percent of participants who actively participate in SMBP monitoring
Costs | During trial; 12 months
  Costs (including time, equipment, consumables) of SMBP monitoring + implementation strategies
Patient Activation | Baseline, 12 months
  Patient Assessment of Chronic Illness Care (PACIC) - Minimum score: 1, Maximum score: 5. The PACIC is scored by summing participants' responses across all 20 items then dividing by 20, the number of items in the scale. Thus, scores on the PACIC range from 1 to 5 with higher scores indicating a better outcome (patient's perception of greater involvement in self-management and receipt of chronic care counseling).

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Khoong, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khoong EC, Kim HC, Li J, Larreynaga J, Luna I, Yang A, Kazi DS, Lyles CR, McCulloch C, Rahman SB, Sarkar U, Curtis N. Implementation Strategies for Self-Measured Blood Pressure Monitoring in Racially and Ethnically Diverse Populations (InSPIRED): A study protocol. Contemp Clin Trials. 2025 Nov;158:108101. doi: 10.1016/j.cct.2025.108101. Epub 2025 Oct 6. PMID 41057081

DOCUMENTS (1):
  • Informed Consent Form (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT06871462/ICF_000.pdf